CLINICAL TRIAL: NCT04414878
Title: A Prospective, Multicenter, Single-arm, Objective Performance Clinical Investigation For Evaluation of the Safety and Effectiveness of MicroPort™ CardioFlow VitaFlow ™ II Transcatheter Aortic Valve System in the Treatment of Severe Aortic Valve Stenosis
Brief Title: VitaFlow™ II Transcatheter Aortic Valve System Pre-market Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort CardioFlow Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUPERIOR-2017
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm clinical investigation (Experimental): Subjects in experimental group will be implanted with the VitaFlow™ II Transcatheter Aortic Valve System
  Interventions: Device: VitaFlow™ II Transcatheter Aortic Valve System

INTERVENTIONS:
Device: VitaFlow™ II Transcatheter Aortic Valve System — VitaFlow™ II Transcatheter Aortic Valve System contains a valve stent-VitaFlow™ Aortic Valve, a delivery system-VitaFlow™ Delivery System, loading tools, and a guide-wire

SUMMARY:
This is a pre-market clinical investigation aiming to evaluate the safety and effectiveness of Microport™ CardioFlow VitaFlow™ II Transcatheter Aortic Valve System for the treatment of severe aortic stenosis.

DETAILED DESCRIPTION:
This a prospective, multi-center, single-arm, objective performance clinical investigation, aiming to evaluate the safety and effectiveness of Microport™ CardioFlow VitaFlow™ II Transcatheter Aortic Valve System for the treatment of severe aortic stenosis. A total of 145 subjects will be enrolled in 18 clinical centers within China. Clinical or telephone follow-up is scheduled at 30 days, 6 months, 12 months, and 2-5 years after valve implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥70 years;
2. Symptomatic , severe, aortic valve stenosis : peak velocity ≥4.0m/s, or mean transvalvular gradient ≥40mmHg(1 mmHg=0.133kPa), or effective orifice area<0.8cm² (or EOA index<0.5cm²/m²);
3. NYHA≥II class;
4. Estimated life-expectancy>12 months after implantation of the prosthetic valve;
5. Anatomically suitable for the transcatheter aortic valve implantation procedure;
6. The patients considered to high-risk or not suitable for surgical aortic valve replacement (SAVR), as assessed by two or above heart surgeons; The patient has been informed of the nature of the study, is willing to enroll in the study by signing a patient informed consent and agreeing to the scheduled follow up requirement.

Exclusion Criteria:

1. Acute myocardial infarction (MI) in last 30 days before the treatment;
2. Aortic root anatomy not suitable for the implantation of the transcatheter aortic valve；
3. Complicated lesion of the aortic valve (aortic stenosis with severe regurgitation); moderate-severe mitral valve stenosis; severe mitral valve regurgitation; severe tricuspid valve regurgitation;
4. Previous implantation of heart valve at any position；
5. Hemodynamic instability requiring mechanical hemodynamic support devices;
6. Need for emergency surgery for any reason;
7. Hypertrophic cardiomyopathy with obstruction;
8. Severe left ventricular dysfunction with left ventricular ejection fraction (LVEF) < 20%;Severe right ventricular dysfunction;
9. Active peptic ulcer or upper gastro-intestinal bleeding within the past 3 months;
10. Known hypersensitivity or contraindication to all anticoagulation/antiplatelet regimens, to nitinol, contrast media or other relevant elements.
11. Congenital aortic valve stenosis or unicuspid aortic valve;
12. Vascular diseases or anatomical condition preventing the device access;
13. Active endocarditis or other active infections at the time of treatment;
14. Participating in another trial and the primary endpoint is not achieved.
15. Inability to comply with the clinical investigation follow-up or other requirements.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Rate of all-cause mortality at 12 months post implantation | 12 months post implantation
  Rate of all-cause mortality including cardiovascular and non-cardiovascular death

SECONDARY OUTCOMES:
Valve function-mean prosthetic valve gradient | at 30 days, 6 months, and 1 year post implantation
  Mean prosthetic valve gradient measured by transthoracic echocardiography (TTE)(in mmHg)
Valve function- effective orifice area | at 30 days, 6 months, and 1 year post implantation
  Effective orifice area measured by transthoracic echocardiography (TTE)(in cm^2)
Valve function- degree of prosthetic valve regurgitation | at 30 days, 6 months, and 1 year post implantation
  Degree of prosthetic valve regurgitation including paravalvular leak and intravalvular regurgitation measured by transthoracic echocardiography (TTE)
Rate of safety events according to VARC2 | at 30 days, 6 months, 1 year and annually up to 5 years post implantation
  Rate of safety events according to VARC2 including all-cause mortality, myocardial infarction, stroke, bleeding, acute kidney injury, vascular complications, conduction disturbance and arrhythmias, and new permanent pacemaker implantation
Rate of other TAVI-related complications | at 30 days, 6 months, 1 year and annually up to 5 years post implantation
  Rate of other TAVI-related complications including conversion to open surgery, unplanned use of cardiopulmonary bypass, coronary obstruction, ventricular septal perforation, mitral valve apparatus damage or dysfunction, cardiac tamponade, endocarditis, valve thrombosis, valve mal-positioning, and TAV-in-TAV
Rate of major adverse cardiac and cerebrovascular events(MACCE) | at 30 days, 6 months, 1 year and annually up to 5 years post implantation
  Rate of MACCE including all-cause mortality, stroke, myocardial infarction, re-intervention, arrhythmias, and conduction disturbances
Rate of device success | at immediate post implantation
  Rate of device success, assessed by death, the access, delivery, deployment and implantation of the device, prosthetic valve position and valve function
Rate of balloon pre-dilation success | at immediate post implantation
  Rate of balloon pre-dilation success, assessed by the access, delivery, pre-dilation and retrieval of the balloon catheter
Rate of balloon post-dilation success | at immediate post implantation
  Rate of balloon post-dilation success, assessed by the access, delivery, post-dilation and retrieval of the balloon catheter
Rate of procedure success | at immediate post implantation
  Rate of procedure success, assessed by the device success and the peri-procedural complications

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Fuwai Hospital, Beijing, Beijing Municipality
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang